CLINICAL TRIAL: NCT00251589
Title: A Phase I/II Clinical Trial of Oral Vorinostat (MK0683) in Combination With Erlotinib in Patients With Relapsed/Refractory Non-Small-Cell Lung Cancer
Brief Title: A Phase I/II Clinical Trial of Vorinostat in Combination With Erlotinib for Patients With Relapsed/Refractory Non-Small-Cell Lung Cancer (0683-025)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This trial is being closed based on lack of substantive efficacy, slow accrual and overall tolerance in patients treated to date.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-025; MK0683-025 (Other: Merck); 2005_080 (Other: Merck)
Record Dates: First submitted 2005-11-07; First posted 2005-11-10 (Estimated); Results first posted 2009-03-10 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Relapsed Non-Small-Cell Lung Cancer; Refractory Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (Experimental): Vorinostat 200 mg twice a day for 3 days a week + erlotinib 150 mg once a day was evaluated in the Phase I portion of the study and determined to be the MTD and therefore the recommended Phase II dose. Of the 16 patients treated at this dose level, 4 were assigned to the Phase I portion of the study and 12 were assigned to the Phase II portion
  Interventions: Drug: Vorinostat; Drug: erlotinib
- Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (Experimental): Vorinostat 300 mg once a day for 3 days a week + erlotinib 150 mg once a day was evaluated in the Phase I portion of the amended study and exceeded the MTD. All patients treated at this dose level were assigned to the Phase I portion of the study.
  Interventions: Drug: Vorinostat; Drug: erlotinib
- Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (Experimental): Vorinostat 300 mg twice a day for 3 days a week + erlotinib 150 mg once a day was evaluated in the Phase I portion of the study and exceeded the MTD. All patients treated at this dose level were assigned to the Phase I portion of the study.
  Interventions: Drug: Vorinostat; Drug: erlotinib
- Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk (Experimental): Vorinostat 400 mg once a day for 21 out of 28 days + erlotinib 150 mg once a day was evaluated in the Phase I portion of the original study and exceeded MTD. This cohort was then amended (Amendment 1) to identify a more tolerable once daily vorinostat dosing regimen. All patients treated at this dose level were assigned to the Phase I portion of the study.
  Interventions: Drug: Vorinostat; Drug: erlotinib

INTERVENTIONS:
Drug: Vorinostat — Vorinostat 200 mg twice a day for 3 days a week.
  Other Names: MK0683; Zolinza®
  Arms: Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk
Drug: Vorinostat — Vorinostat 300 mg once a day for 3 days a week.
  Other Names: MK0683; Zolinza®
  Arms: Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk
Drug: Vorinostat — Vorinostat 300 mg twice a day for 3 days a week.
  Other Names: MK0683; Zolinza®
  Arms: Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk
Drug: Vorinostat — Vorinostat 400 mg once a day for 21 out of 28 days.
  Other Names: MK0683; Zolinza®
  Arms: Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Drug: erlotinib — erlotinib 150 mg once a day.
  Other Names: Tarceva ®

SUMMARY:
The reason for this study will be to find the safest maximum tolerated dose of oral vorinostat in combination with erlotinib [Tarceva (TM)] that can be given to patients with lung cancer who have relapsed or failed other therapy for the disease. Once the safest maximum tolerated dose of vorinostat is determined, patients enrolled in the clinical trial will continue vorinostat and erlotinib for up to 8 months. Safety and effectiveness will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age and older with a confirmed diagnosis of non-small-cell lung cancer (NSCLC) who have failed at least one prior treatment for NSCLC.
* Patients must have proven disease by CT scan or MRI.
* Patients must be at least 4 weeks from any chemotherapy for cancer or from any surgeries or from any treatment using an investigational drug.
* Patients must be 2 weeks out from radiation therapy.
* At screening the patient must have normal lab results and can not be pregnant.
* Women and men must agree to practice adequate birth control during the study.
* Patient has the ability to understand and sign the consent form.

Exclusion Criteria:

* Patient had prior treatment with vorinostat or erlotinib.
* Patient has any of the following conditions: active infections including hepatitis B or C, unstable brain metastases, swallowing difficulties, heart problems, significant eye abnormalities, drug or alcohol abuse, mental illness or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 12 investigative sites in the United States. The first patient's first visit was 30 March 2006. The study was terminated early on 12 Oct 2007 and the last patient's last visit was 30 Oct 2007.
Pre-assignment Details: Enrolled patients were assigned to 1 of 2 dose escalating cohorts (A and B) in the Phase I portion of the study to determine the maximum tolerated dose (MTD). Once determined, new patients were assigned to the Phase II portion of the study and treated with the MTD. Active Phase I patients continued into Phase II.
Period: Overall Study
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Started | 16 (4 of the 16 patients participated in Phase I and II portions. 12 participated in Phase II only.) | 3 | 2 | 2
Completed | 1 | 0 | 0 | 0
Not Completed | 15 | 3 | 2 | 2
Not completed — Adverse Event | 5 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Discontinued due to progressive disease | 9 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk | Total
Number analyzed (Participants) | 16 | 3 | 2 | 2 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (4.36) | 66.0 (8.49) | 48.5 (20.51) | 59.1 (11.59) | 60.7 (11.41)
Age, Customized [Number; unit: Participants]
  ≤ 65 years | 11 | 3 | 1 | 2 | 17
  > 65 years | 5 | 0 | 1 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 1 | 1 | 12
  Male | 8 | 1 | 1 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) Occurring in Cycle 1 of the Phase I Portion of the Study
Description: Adverse event(s) that determined the treatment dose level was not tolerable for that patient in Cycle 1 of the Phase I portion of the study.
Time Frame: Day 1 to 28 in the Phase I portion of the study
Population: All patients as treated population in Cycle 1 of the Phase I portion of the study.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 4 | 3 | 2 | 2
Participants | 0 | 2 | 2 | 1

2. Secondary Outcome: Unconfirmed Partial Response (UPR) Based on Response Criteria in Solid Tumors (RECIST)
Description: An unconfirmed partial response is defined as a partial response that has not been confirmed by a follow up CT scan (or MRI) at least 4 weeks after the criteria for response are first met. (A partial response is defined as an at least 30% reduction in the sum of the longest diameter of the target lesions. Non-target lesions must be at least stable)
Time Frame: Every 57 days beginning with Cycle 3, or more frequently if appropriate
Population: All patients as treated population with post-baseline data available to determine Unconfirmed Partial Response as Best Response.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 13 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Dose Limiting Toxicity Occurring in Cycle 1 of the Phase II Portion of the Study
Description: Adverse event(s) that determined the treatment dose level was not tolerable for that patient in Cycle 1 of the Phase II portion of the study.
Time Frame: Day 1 to 28 in the Phase II portion of the study
Population: All patients as treated population in Cycle 1 of the Phase II portion of the study.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 12 | 0 | 0 | 0
Participants | 3 |  |  |

4. Post Hoc Outcome: Dose Limiting Toxicity Occurring in Cycles 2 and Beyond of the Phase II Portion of the Study
Description: Adverse event(s) that determined the treatment dose level was not tolerable for that patient in Cycles 2 and beyond of the Phase II portion of the study.
Time Frame: After day 28 in the Phase II portion of the study
Population: All patients as treated population in Cycles 2 and beyond of the Phase II portion of the study.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 12 | 0 | 0 | 0
Participants | 3 |  |  |

5. Secondary Outcome: Stable Disease (SD) as Best Response Based on Response Criteria in Solid Tumors (RECIST)
Description: Stable disease is defined as less than a radiographic partial response, but not progressive disease
Time Frame: Every 57 days beginning with Cycle 3, or more frequently if appropriate
Population: All patients treated population with post-baseline data available to determine Stable Disease as Best Response.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 13 | 1 | 1 | 1
Participants | 6 | 1 | 1 | 1

6. Secondary Outcome: Progressive Disease (PD) as Best Response Based on Response Criteria in Solid Tumors (RECIST)
Description: Progressive disease is defined as a ≥20% increase in the sum of the longest diameter, the appearance of one or more new lesions and/or unequivocal progression of non-target lesions by conventional or spiral CT or MRI
Time Frame: Every 57 days beginning with Cycle 3, or more frequently if appropriate
Population: All patients as treated population with post-baseline data available to determine Progressive Disease as Best Response.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 13 | 1 | 1 | 1
Participants | 7 | 0 | 0 | 0

7. Secondary Outcome: Disease Progression After Week 8 Based on Response Criteria in Solid Tumors (RECIST)
Description: First documentation of Progressive Disease (PD) occurring > 8 weeks on study.
Time Frame: Every 57 days beginning with Cycle 3 (Week 8), or more frequently if appropriate
Population: All patients as treated population with post-baseline data available to determine Disease Progression After Week 8.
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 13 | 1 | 1 | 1
Participants | 3 | 0 | 0 | 0

8. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was measured from the start of the treatment to the time when the criteria for progression was met or death due to any cause (whichever is first recorded).
Time Frame: Day 1 to disease progression or death
Population: All patients as treated population with post-baseline data available to determine progression free survival.
  Cohort A, Dose Level 1 (Amended), Cohort B, Dose Level 2 and Cohort A, Dose Level 1 (Original) are not represented in the below table as post-baseline data were not available to determine progression free survival.
Measure: Mean (Full Range); unit: Days
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk
Number analyzed (Participants) | 13
Days | 57 [26 to 113]

ADVERSE EVENTS:
Arm/Group | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk
Serious Adverse Events (participants affected / at risk) | 6/16 | 2/3 | 2/2 | 1/2
Other Adverse Events (participants affected / at risk) | 16/16 | 3/3 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (N=16) | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (N=3) | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (N=2) | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk (N=2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 200 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (N=16) | Vorinostat 300 mg q.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (N=3) | Vorinostat 300 mg b.i.d. 3d/wk + Erlotinib 150 mg q.d. 7d/wk (N=2) | Vorinostat 400 mg q.d. 21d/4wk + Erlotinib 150 mg q.d. 7d/wk (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Keratoconjunctivitis sicca (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 13 (32) | 3 (6) | 2 (8) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (21) | 2 (2) | 2 (5) | 2 (3)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (14) | 1 (1) | 2 (3) | 2 (3)
Asthenia (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (14) | 1 (4) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood glucose decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 6 (7) | 1 (2) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 10 (15) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 1 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 9 (13) | 3 (4) | 0 (0) | 2 (6)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the slow pace of patient accrual, failure to observe meaningful efficacy in treated patients, and overall intolerance of the combination regimen, the study was terminated prematurely on 12-Oct-2007.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.